CLINICAL TRIAL: NCT02715349
Title: Psychoeducation for Vietnamese Families With a Patient With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danang Psychiatric Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DPH20140818
Record Dates: First submitted 2016-03-03; First posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Schizophrenia
Keywords: schizophrenia; psychoeducation; Vietnam
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychoeducation (Experimental): 3 session psychoeducation program with the family, and 3 session psychoeducation program with the patient, after psychosis is controlled. Psychoeducation focuses on explaining schizophrenia as a medical illness, the prognosis, and how the patient and family can increase the likelihood of better outcome.
  Interventions: Behavioral: Psychoeducation
- Control (No Intervention): Family and patient do not receive psychoeducation, but still receive standard hospital services for schizophrenia.

INTERVENTIONS:
Behavioral: Psychoeducation — 3 session psychoeducation program with the family, and 3 session psychoeducation program with the patient, after psychosis is controlled. Psychoeducation focuses on explaining schizophrenia as a medical illness, the prognosis, and how the patient and family can increase the likelihood of better outcome.
  Arms: Psychoeducation

SUMMARY:
Families with a patient with schizophrenia and the patient are randomly assigned to receive either a 3 session psychoeducation program, or no psychoeducation. Other treatment for schizophrenia and other mental illness are provided as usual.

DETAILED DESCRIPTION:
Families with a patient with schizophrenia and the patient are randomly assigned to receive either a 3 session psychoeducation program, or no psychoeducation. Other treatment for schizophrenia and other mental illness are provided as usual. The psychoeducation program focuses on: (a) explaining schizophrenia as a medical, biological illness, (b) the prognosis for schizophrenia (e.g., that it is possible to lead a normal life), and (c) what the family and patient can do to maximize the outcome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia, based on ICD-10
* Receive in-patient treatment at hospital
* Length of schizophrenia less than 3 years.
* Treated 3 or less times for schizophrenia.

Exclusion Criteria:

* Mental retardation, or other diagnoses that could affect the ability to answer questionnaires, after the acute schizophrenia psychosis is controlled.
* Suicidal ideation

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline (pre-treatment) to 6 months post-baseline in patient-report of quality of life using the Quality of Life Enjoyment and Satisfaction Questionnaire. | baseline (pre-treatment). six months post-baseline.
  Change in quality of life using an Analysis of Covariance with the baseline quality of life score as the covariate, the 6 month quality of life assessment as the dependent variable, and treatment group as the independent variable. The Quality of Life Enjoyment and Satisfaction Questionnaire with patient-report is used at both timepoints.
Change from baseline (pre-treatment) at 6 months post-baseline in family-report of quality of life using the Quality of Life Enjoyment and Satisfaction Questionnaire. | baseline (pre-treatment). six months post-baseline.
  Change in quality of life using an Analysis of Covariance with the baseline quality of life score as the covariate, the 6 month quality of life assessment as the dependent variable, and treatment group as the independent variable. The Quality of Life Enjoyment and Satisfaction Questionnaire with family-report is used at both timepoints.

SECONDARY OUTCOMES:
Change from baseline (pre-treatment) to 6 months post-baseline in patient-report of stigma towards schizophrenia using the Stigma Towards Schizophrenia questionnaire. | baseline (pre-treatment). six months post-baseline.
  Change in stigma towards schizophrenia using an Analysis of Covariance with the baseline stigma towards schizophrenia as the covariate, the 6 month stigma towards schizophrenia assessment as the dependent variable, and treatment group as the independent variable. The Stigma Towards Schizophrenia with patient-report is used at both timepoints.
Change from baseline (pre-treatment) to 6 months post-baseline in family-report of stigma towards schizophrenia using the Stigma Towards Schizophrenia questionnaire. | baseline (pre-treatment). six months post-baseline.
  Change in stigma towards schizophrenia using an Analysis of Covariance with the baseline stigma towards schizophrenia as the covariate, the 6 month stigma towards schizophrenia assessment as the dependent variable, and treatment group as the independent variable. The Stigma Towards Schizophrenia with family-report is used at both timepoints.
Patient-report for schizophrenia medication compliance, at 6 months post-baseline | 6 months post-baseline
  Analysis of Variance on medication compliance as reported by the patient

OTHER OUTCOMES:
Patient-report satisfaction with hospital services, at 6 months post-baseline | 6 months post-baseline
  Patient-report satisfaction with services provided by the hospital.
Family-report satisfaction with hospital services, at 6 months post-baseline | 6 months post-baseline
  Family-report satisfaction with services provided by the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Ngoc Tran, MD, Principal Investigator — Danang Psychiatric Hospital
Locations (1):
- Danang Psychiatric Hospital, Da Nang, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided